CLINICAL TRIAL: NCT04399993
Title: Effect of Osteopathic Manual Techniques on the Diaphragm Muscle and Its Repercussions in Healthy Young Adults
Brief Title: Effect of Osteopathic Manual Techniques on the Diaphragm Muscle and Its Repercussions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OST1- 001
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Osteopathy; Diaphragm; Center of Pressure; Range of Motion; Thoracolumbar
MeSH Terms: interventions — Contraceptive Devices, Female

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The volunteers will be allocated randomly using a website called radom.org, which ensures that neither neither the volunteer nor the assessor will know the final allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Protocol in Diaphragm (Experimental): In each volunteer, after a brief questionnaire, it will be measured the center of gravity and the range of movement of the lumbar spine before the technique.
  Each volunteer will stay in supine position with arms along their body, in which their legs may be either extended or flexed.
  Next, the researcher will perform the intervention protocol in Diaphragm. Then, all the measurements described before, will be repeated by the assessor right after the technique.
  Interventions: Other: Intervention Protocol in Diaphragm
- Sham Technique (Sham Comparator): In each volunteer, after a brief questionnaire, it will be measured the center of gravity and the range of movement of the lumbar spine before the technique.
  Each volunteer will stay in supine position with arms along their body, in which their legs may be either extended or flexed.
  Next, the researcher will perform the Sham technique. Then, all the measurements described before, will be repeated by the assessor right after the technique.
  Interventions: Other: Sham technique

INTERVENTIONS:
Other: Intervention Protocol in Diaphragm — The protocol consists of three techniques. The two first techniques will be applied for 10 respiratory cycles.
  Muscle Stretching Technique:
  the researcher will perform a cephalic traction on the inferior costal border with the ulnar border during the inspiratory phase.
  Phrenic-center inhibition technique:
  the researcher, with a hand on the sternum to caudal and other hand on the umbilical region to cranial, will approach his hands on the horizontal plane, when the volunteer exales.
  Functional diaphragm technique:
  the researcher will perform a vertical pressure on the diaphragm for 5 minutes and will search for the facilitated parameters and maintain them until the release of all the periarticular elements.
  Arms: Intervention Protocol in Diaphragm
Other: Sham technique — In the sham group a manual contact without any therapeutic intention will be performed, in a distant region of the diaphragm (for example on the trapezius muscle). This contact will be maintained during the same amount of time as for the treatment group.
  Arms: Sham Technique

SUMMARY:
Determining the effects of an intervention plan on the diaphragm related to the center of gravity and range of motion in the lumbar spine (static and dynamic) in healthy individuals is an area that lacks evidence and proper studies. Has such, the investigators consider this a interesting topic to study, therefore it is intended to improve the knowledge on this area.

DETAILED DESCRIPTION:
All diaphragmatic activity is controlled by metabolic mechanisms and emotional states which may cause restrictions that might be related to disorders in the lower back.

The diaphragm and the lumbar segment of the spine are connected through the diaphgramathic pillars that connect the central tendon and the vertebrae of L2 (left side) and L3/L4 (right side). Consequently, the contraction of the pillars may be related to the fixation of the lumbar spine.

Proper function of the diaphragm is related to better parameters of static balance. It is also possible to conclude that a change in the proper function of the diaphragm is associated with changes in the center of gravity in healthy individuals.

This theme lacks scientific evidence, since no studies were found that focus on the analysis of diaphragmatic treatment only. In this way, the investigators intend to collaborate to increase knowledge in this area, determining the effects of the intervention plan on the diaphragm in relation to the range of motion and center of gravity in the lumbar spine (static and dynamic) in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 30 years old;
* Both genders;

Exclusion Criteria:

* Treatments with manual therapy in the last three months or more than three times in the previous year;
* Lumbar spine pathology (infection, spinal fracture or more severe neurological impairment, such as cauda equina syndrome) and respiratory pathologies;
* Psychiatric illness;
* Recent history of trauma;
* History of cancer;
* Systemic inflammatory conditions;
* Recent history of spinal surgery;
* Abdominal pain at the time of the intervention;
* Body mass index (BMI) equal to or greater than 31kg / m2, due to the difficulty in accessing the diaphragm;
* All of those that acquired a higher knowledge within the area of manual therapy, which may compromise its validation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of Center of gravity immediately after the intervention | Immediately after the intervention
  To obtain the center of gravity measurements, it will be used the system Qualisys Track Manager. First, it will be placed in the subject spheric markers on the spinous processes of T12, L3 and S2 and both anterior and posterior superior iliac spines.
  The cameras will be arranged to cover the area to the test, which it will be performed in a hard surface with the help of reflector-markers that will evaluate the movements.
  The data will be collected twice, with the eyes open and closed. They'll be standing in the platform for 90 seconds each time and the data will be collected at the 30, 60 and 90 seconds.
  The software is going to be used to convert the data in coordinates in the x, y and z axis, which it will allow to analyse the tridimensional kinematics of the lumbar spine Through the intrinsical board of Qualysis Track Manager it will be evaluated the relation of the center of pressure with the vertical projection of the center of mass through the distance between both.

SECONDARY OUTCOMES:
Change from Baseline in Range of Movement of the lumbar spine immediately after the intervention | Immediately after the intervention
  To obtain the center of gravity measurements, it will be used the system Qualisys Track Manager. First, it will be placed in the subject spheric markers on the spinous processes of T12, L3 and S2 and both anterior and posterior superior iliac spines.
  The cameras will be arranged to cover the area to the test, which it will be performed in a hard surface with the help of reflector-markers that will evaluate the movements.
  The data will be collected by asking the volunteer to perform certain movements such as anterior and lateral flexion.
  The software is going to be used to convert the data in coordinates in the x, y and z axis, which it will allow to analyse the tridimensional kinematics of the lumbar spine Through the intrinsical board of Qualysis Track Manager it will be evaluated the relation of the center of pressure with the vertical projection of the center of mass through the distance between both.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Saúde do Politécnico do Porto
Locations (1):
- Escola Superior de Saúde do Politécnico do Porto, Porto, Portugal

REFERENCES:
- [Background] Licciardone JC, Kearns CM, Minotti DE. Outcomes of osteopathic manual treatment for chronic low back pain according to baseline pain severity: results from the OSTEOPATHIC Trial. Man Ther. 2013 Dec;18(6):533-40. doi: 10.1016/j.math.2013.05.006. Epub 2013 Jun 10. PMID 23759340
- [Background] Acute low back problems in adults: assessment and treatment. Agency for Health Care Policy and Research. Clin Pract Guidel Quick Ref Guide Clin. 1994 Dec;(14):iii-iv, 1-25. PMID 7987418
- [Background] Nason LK, Walker CM, McNeeley MF, Burivong W, Fligner CL, Godwin JD. Imaging of the diaphragm: anatomy and function. Radiographics. 2012 Mar-Apr;32(2):E51-70. doi: 10.1148/rg.322115127. PMID 22411950
- [Background] Grams ST, von Saltiel R, Mayer AF, Schivinski CI, de S Nobre LF, Nobrega IS, Jacomino ME, Paulin E. Assessment of the reproducibility of the indirect ultrasound method of measuring diaphragm mobility. Clin Physiol Funct Imaging. 2014 Jan;34(1):18-25. doi: 10.1111/cpf.12058. Epub 2013 Jun 4. PMID 23730805
- [Background] van Tulder M, Becker A, Bekkering T, Breen A, del Real MT, Hutchinson A, Koes B, Laerum E, Malmivaara A; COST B13 Working Group on Guidelines for the Management of Acute Low Back Pain in Primary Care. Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S169-91. doi: 10.1007/s00586-006-1071-2. No abstract available. PMID 16550447
- [Background] Marti-Salvador M, Hidalgo-Moreno L, Domenech-Fernandez J, Lison JF, Arguisuelas MD. Osteopathic Manipulative Treatment Including Specific Diaphragm Techniques Improves Pain and Disability in Chronic Nonspecific Low Back Pain: A Randomized Trial. Arch Phys Med Rehabil. 2018 Sep;99(9):1720-1729. doi: 10.1016/j.apmr.2018.04.022. Epub 2018 May 19. PMID 29787734
- [Background] Savigny P, Watson P, Underwood M; Guideline Development Group. Early management of persistent non-specific low back pain: summary of NICE guidance. BMJ. 2009 Jun 4;338:b1805. doi: 10.1136/bmj.b1805. No abstract available. PMID 19502217
- [Background] Rubinstein SM, van Middelkoop M, Assendelft WJ, de Boer MR, van Tulder MW. Spinal manipulative therapy for chronic low-back pain: an update of a Cochrane review. Spine (Phila Pa 1976). 2011 Jun;36(13):E825-46. doi: 10.1097/BRS.0b013e3182197fe1. PMID 21593658
- [Background] Hagg O, Fritzell P, Nordwall A; Swedish Lumbar Spine Study Group. The clinical importance of changes in outcome scores after treatment for chronic low back pain. Eur Spine J. 2003 Feb;12(1):12-20. doi: 10.1007/s00586-002-0464-0. Epub 2002 Oct 24. PMID 12592542
- [Background] Bagheri R, Ebrahimi Takamjani I, Dadgoo M, Ahmadi A, Sarrafzadeh J, Pourahmadi MR, Jafarpisheh AS. Gender-Related Differences in Reliability of Thorax, Lumbar, and Pelvis Kinematics During Gait in Patients With Non-specific Chronic Low Back Pain. Ann Rehabil Med. 2018 Apr;42(2):239-249. doi: 10.5535/arm.2018.42.2.239. Epub 2018 Apr 30. PMID 29765877
- [Background] Shahbazi Moheb Seraj M, Sarrafzadeh J, Maroufi N, Ebrahimi Takamjani I, Ahmadi A, Negahban H. The Ratio of Lumbar to Hip Motion during the Trunk Flexion in Patients with Mechanical Chronic Low Back Pain According to O'Sullivan Classification System: A Cross-sectional Study. Arch Bone Jt Surg. 2018 Nov;6(6):560-569. PMID 30637313
- [Background] Wu G, Siegler S, Allard P, Kirtley C, Leardini A, Rosenbaum D, Whittle M, D'Lima DD, Cristofolini L, Witte H, Schmid O, Stokes I; Standardization and Terminology Committee of the International Society of Biomechanics. ISB recommendation on definitions of joint coordinate system of various joints for the reporting of human joint motion--part I: ankle, hip, and spine. International Society of Biomechanics. J Biomech. 2002 Apr;35(4):543-8. doi: 10.1016/s0021-9290(01)00222-6. PMID 11934426
- [Background] Masani K, Vette AH, Kouzaki M, Kanehisa H, Fukunaga T, Popovic MR. Larger center of pressure minus center of gravity in the elderly induces larger body acceleration during quiet standing. Neurosci Lett. 2007 Jul 18;422(3):202-6. doi: 10.1016/j.neulet.2007.06.019. Epub 2007 Jun 17. PMID 17611029
- [Background] Doyle RJ, Hsiao-Wecksler ET, Ragan BG, Rosengren KS. Generalizability of center of pressure measures of quiet standing. Gait Posture. 2007 Feb;25(2):166-71. doi: 10.1016/j.gaitpost.2006.03.004. Epub 2006 Apr 19. PMID 16624560
- [Background] Qualisys, A. B., & Gothenburg, S. (2011). Qualisys track manager. New York: User Manual.
- [Background] Zemková, E. (2011). Assessment of balance in sport: Science and reality. Serbian Journal of Sports Sciences, (4).
- [Background] Donlon, T., Franklin, B., Machamer, C., Mogelnicki, C., Verneus, J., & Taber, C. (2018). FMS Squat Assessment and 2D Video Motion Analysis as Screening Indicators of Low Back Pain: A Cross Sectional Case-Study.
- [Background] Souchard, P. E. (1989). O diafragma. Summus editorial.